CLINICAL TRIAL: NCT06521112
Title: The Effect of Oral Care on Mucositis and Oral Mucosa in Intensive Care Unit Patients According to Individual Oral Care Frequency Assessment
Brief Title: The Effect of Oral Care on Mucositis and Oral Mucosa According to Individual Oral Care Frequency Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ülkü özdemir, associate professor doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YS2022
Record Dates: First submitted 2024-07-08; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mucositis
Keywords: Intensive care unit; Oral care; Nursing; Oral mucosa; Mucositis
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Intervention Model Description: a randomized, controlled trial in pre-test post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Individual daily oral care frequency will not be determined for each patient in the control group.
  0.2% chlorhexidine for 2 minutes, once per shift as frequently as the clinic routinely applies (3 shifts in total: once between 08:00-16:00; 16:00-24:00; 24:00-08:00) standard oral care will be applied with the solution containing.
- Intervention Group (Experimental): Morning shift every day for 10 days; An individual Intensive Care Oral Care Frequency Rating Scale will be applied to each patient daily.
  According to the results of the Intensive Care Oral Care Frequency Evaluation Scale, individual oral care frequency will be planned for each patient daily and recorded in the patient follow-up form.
  Then, oral care will be applied with a solution containing 0.2% chlorhexidine gluconate for 2 minutes, in line with the clinical protocol and at the planned frequency.
  Interventions: Drug: Oral care with a solution containing 0.2% chlorhexidine gluconate a frequency determined according to the results of the Intensive Care Oral Care Frequency Rating Scale.

INTERVENTIONS:
Drug: Oral care with a solution containing 0.2% chlorhexidine gluconate a frequency determined according to the results of the Intensive Care Oral Care Frequency Rating Scale. — Every day for 10 days, Frequency determined according to Intensive Care Oral Care Frequency Rating Scale, Oral care was applied for 2 minutes a solution containing 0.2% chlorhexidine gluconate.
  Other Names: KARYA
  Arms: Intervention Group

SUMMARY:
The aim of the study is to examine the effect of oral care based on individual oral care frequency assessment on mucositis and oral mucosa integrity in intensive care patients, instead of standard routine oral care practice.

The study was planned as a randomized controlled experimental study. The population of the research consists of patients hospitalized in the Internal Medicine Intensive Care Unit of Erciyes University Health Application and Research Center in Kayseri. In determining the groups, randomization was planned to be determined by lottery method, and patients were assigned to groups with odd and even bed numbers accordingly. In the study, data were collected using the Patient Information Form, Intensive Care Oral Care Frequency Assessment Scale, World Health Organization Mucositis Evaluation Form and Patient Follow-up Form.

DETAILED DESCRIPTION:
The research was conducted as a randomized, observational drug study to examine the effect of oral care based on individual oral care frequency assessment on mucositis and oral mucosal integrity in intensive care patients, instead of standard oral care practice. Intervention and control groups were used in the study. While performing oral care, which forms the basis of the study, support was received from intensive care nurses with experience in accordance with the procedure steps.

The population of the research consists of patients hospitalized in the Internal Medicine Intensive Care Unit of Erciyes University Health Application and Research Center.

For the sample size, 21-20 patients were included in the control and intervention groups, respectively, between May 2023 and December 2023.

In the assignment of groups, randomization was planned to be determined by lottery method, and accordingly, patients were assigned to groups with odd bed numbers and even bed numbers. From time to time, patient beds were closed (due to lack of personnel) and no patient admissions could be made. In this case, there could be differences in the characteristics of the patients who could be admitted to each bed. Equivalence of the groups in terms of age, gender and disease characteristics was ensured by randomization.

Applications to the Intervention Group Patients in the intervention group were administered the Patient Information Form, Intensive Care Oral Care Frequency Evaluation Scale, World Health Organization Mucositis Evaluation Form and Oral Evaluation Guide on the first day. Oral care frequency was planned according to the results of the oral care frequency assessment scale. The measurements taken and the planned oral care frequency were recorded in the patient follow-up form. Then, oral care was given at the planned frequency in line with the clinical protocol and according to the results of the Oral Care Frequency Evaluation Scale. Oral care starts with creating a suitable environment; The patient's mouth care swabs were prepared by wetting them with a solution (containing 0.2% chlorhexidine gluconate) for each application, 4 equal to each patient. If the patient was conscious, he was given a comfortable position. If he was not conscious, the patient's head was turned towards the person who will perform the procedure. The patient was kept in a side-lying position, and oral care was given to the patient, covering the patient's teeth, inner cheeks, sublingual, gums and all other soft tissues. After the patient's oral care procedure was completed, the procedure was terminated by giving the patient his previous position. Each treatment lasted no less than 2 minutes (min.).

Then, the Intensive Care Oral Frequency Evaluation Scale, World Health Organization Mucositis Evaluation Form and Oral Evaluation Guide were applied every morning shift for 10 days, and daily oral care frequency was planned according to the results of the oral care frequency evaluation scale. The measurements taken and the planned oral care frequency were recorded in the patient follow-up form. Then, oral care was given in accordance with the clinical protocol and at the determined frequency.

After the tenth day was completed, the World Health Organization Mucositis Evaluation Form and Oral Evaluation Guide were applied again.

Oral care will be performed with the solution currently used by the clinic, and existing application solutions will not be interfered with. The study was terminated for patients whose oral care solutions were changed during the study.

Applications to the Control Group Patients in the control group were administered the Patient Information Form, World Health Organization Mucositis Evaluation Form and Oral Evaluation Guide on the first day. Then, oral care was given at the frequency of the clinic's routine and in line with the clinic protocol. The daily oral care routine of the clinic was applied once per shift (there are 3 shifts in total; 08:00-16:00; 16:00-24:00; 24:00-08:00) as a standard. Oral care starts with creating a suitable environment; The patient's mouth care swabs were prepared by wetting them with a solution (containing 0.2% chlorhexidine gluconate) for each application, 4 equal to each patient. If the patient was conscious, he was given a comfortable position. If he was not conscious, the patient's head was turned towards the person who will perform the procedure. The patient was kept in a side-lying position, and oral care was given to the patient, covering the patient's teeth, inner cheeks, sublingual, gums and all other soft tissues. After the patient's oral care procedure was completed, the procedure was terminated by giving the patient his previous position. Each treatment lasted no less than 2 minutes (min.).

Then, the World Health Organization Mucositis Evaluation Form and Oral Evaluation Guide were applied every morning shift for 10 days, and the measurements and the routine oral care frequency of the clinic were recorded on the patient follow-up form. Then, oral care was given at the clinic's routine frequency and in line with the clinic protocol.

After the tenth day was completed, the World Health Organization Mucositis Evaluation Form and Oral Evaluation Guide were again in compliance.

Oral care will be performed with the solutions currently used by the clinic, and existing application solutions will not be interfered with. The study was terminated for patients whose oral care solutions were changed during the study.

The suitability of the data for normal distribution was evaluated with histogram, Q-Q graphs and Shapiro-wilk test. Homogeneity of variance was tested with the Levene test. In comparisons between groups, independent two-sample t-test was applied for quantitative variables. One-way analysis of variance was used for comparisons between more than two groups. Paired t test was used for quantitative variables in repeated pairwise comparisons. . Comparisons between more than two repeated measurements were evaluated by analysis of variance in repeated measurements. Pearson χ2 analysis and Fisher exact χ2 test were used for comparisons of categorical data. Bonferroni, Tukey and Tamhane tests were applied for multiple comparisons. The significance level was accepted as p<0.05.

Ethics committee approval (decision no: 2022/751) from the Erciyes University Clinical Research Ethics Committee and written permission from the unit where the study would be conducted were obtained in order to conduct the study. In addition, those whose written consent was obtained through the Informed Consent Form were included in the study.

ELIGIBILITY:
Inclusion Criteria;

1. Patients aged 18 and over,
2. Patients in the Internal Medicine Intensive Care Unit,
3. According to the World Health Organization Mucositis Evaluation Form, patients who do not have mucositis and patients who have mucositis but do not require additional treatment,
4. Conscious patients/relatives of unconscious patients who agreed to participate in the study and whose voluntary consent was obtained,
5. Patients who are not allergic to the oral care solution or mouthwash ingredients to be used will be included in the study.

Exclusion Criteria;

1. Patients under the age of 18,
2. Patients who do not accept the study,
3. Patients who are allergic to the oral care solution or mouthwash ingredients to be used,
4. Patient groups who have operations in the mouth and for whom oral care is contraindicated,
5. Patients with head and neck cancer receiving radiotherapy will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
World Health Organization Mucositis Evaluation Form | eleven days
  World Health Organization Oral Mucositis Evaluation Form is used in healthcare institutions to evaluate the oral mucosa and determine the degree of oral mucositis. . According to this form, mucositis degrees are scored between 0 and 4 points. While performing this scoring, the oral mucosa of individuals is evaluated both objectively (erythema, ulceration, etc.), subjectively (oral pain, etc.) and functionally (patient's ability to eat, etc.). These ratings; 0: no oral mucositis; 1 point is mild; 2 points is medium; 3 points are serious; A score of 4 indicates the presence of life-threatening mucositis.
Oral Evaluation Guide | eleven days
  The Oral Evaluation Guide, which is a frequently used guide in our country, was created by Eilers et al. in 1988. The guide consists of 8 headings. The titles are examined to provide information about individuals' oral and dental health. These titles; condition of voice, swallowing, lips, tongue, saliva, mucous membranes, gums, teeth or dentures. Each variable is prepared to receive 1, 2 or 3 points, and the dialect evaluation score is obtained by summing these points. A minimum of 8 and a maximum of 24 points can be obtained in the guide. In line with the guide, low scores indicate that the oral mucosa health is good, while high scores indicate that the oral mucosal health is poor.
Intensive Care Oral Care Frequency Rating Scale | ten day
  The scale includes nine parameters. These; It consists of the following topics: age, lips, teeth, tongue, oral mucosa, saliva, cheeks, nutritional support and respiratory support. Each parameter is evaluated separately as Normal = 1 point, Mild = 2 points, Moderate = 3 points and Severe = 4 points. In cases of broad-spectrum antibiotic or steroid treatment, diabetes mellitus diagnosis, low hemoglobin (Hb) concentration and immunosuppressive drug use, 1 additional point is added to the total score for each condition. According to the total score, the patient's oral care frequency is revealed.

CONTACTS AND LOCATIONS:
Overall Officials: yasar sahin, Principal Investigator — TC Erciyes University; Ülkü Özdemir, Principal Investigator — TC Erciyes University; Recep Civan Yüksel, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No